CLINICAL TRIAL: NCT05997550
Title: The Effect of Pursed Lip Breathing Exercise and Laughter Therapy on Dyspnea, Health Status, and Care Dependence in Individuals With Chronic Obstructive Pulmonary Disease
Brief Title: The Effect of Pursed Lip Breathing Exercise and Laughter Therapy Individuals With The COPD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yuksek Ihtisas University (Other)
Responsible Party: Principal Investigator, Goncagul Aldan, lecturer, Yuksek Ihtisas University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: COPD.NURSİNG.YUKSEK
Record Dates: First submitted 2023-06-16; First posted 2023-08-18 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: Chronic Obstructive Pulmonary Disease; Dyspnea; Health Status; Pursed Lip Breathing Exercise; Laughter Therapy; care Dependence
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Dyspnea | interventions — Laughter Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Pursed Lip Breathing Exercise Group (Active Comparator): During the first interview, the training and demonstration of pursed lip breathing exercise is performed by the thesis student in a single session. After this information session, the pursed lip breathing exercise taught from the patients; They are asked to do it in their own homes, 3 days a week on Monday, Wednesday and Friday, for about 30 minutes each session, for a total of eight weeks. In addition, one day a week (on a day determined by the patient, Monday, Wednesday or Friday), the thesis student makes a video call to the patient on WhatsApp, and the practice of pursed lip breathing exercise is performed during the video call.
  Interventions: Other: Pursed Lip Breathing Exercise
- Laughter Therapy Group (Active Comparator): During the first interview, laughter therapy training and demonstration is carried out by the thesis student in a single session. After this information session, the laughter therapy taught from the patients; They are asked to do this in their own homes, 3 days a week on Monday, Wednesday and Friday, 30 minutes each session, for a total of eight weeks. . In addition, once a week (on a day determined by the patient, Monday, Wednesday or Friday), the thesis student makes a video call to the patient on WhatsApp, and laughter therapy is practiced during the video call.
  Interventions: Other: Laughter Therapy
- Control Group (Placebo Comparator): Attention-match training is given to the patients in the control group. During the first interview, attention matching training is carried out by the thesis student for one time, about "Lung structure and functioning", lasting approximately 20 minutes. In addition, a brochure about lung structure and functioning is given to patients. The patients in the control group are not subjected to any other interventions throughout the study.
  Interventions: Other: the control group.

INTERVENTIONS:
Other: Pursed Lip Breathing Exercise — Pursed Lip Breathing Exercise for The COPD
  Arms: Pursed Lip Breathing Exercise Group
Other: Laughter Therapy — Laughter Therapy for the COPD
  Arms: Laughter Therapy Group
Other: the control group. — Attention-match training is given to the patients in the control group.
  Arms: Control Group

SUMMARY:
Chronic Obstructive Pulmonary Disease is a chronic disease with increasing mortality, morbidity and prevalence in the world and in our country, and in which serious symptoms, especially dyspnea, develop. Due to dyspnea and symptoms, patients experience deterioration in their health status and an increase in care dependency. This research is a single-blind, randomized controlled experimental study designed to determine the effects of pursed lip breathing exercise and laughter therapy on dyspnea severity, health status and care dependence in individuals with COPD. The research will be carried out with a total of 63 patients in Ankara City Hospital Chest Diseases unit. The patients will be stratified according to smoking status and COPD Assessment Test scores with the randomization program and assigned to 2 intervention groups and 1 control group. During the first interview, patients in the 1st intervention group will be provided with pursed lip breathing exercise training and application, and training videos and brochures will be given. 2. The patients in the intervention group will be given laughter therapy training and practice, and an educational brochure will be given. The patients in the control group will also receive face-to-face training on lung structure and functioning, and a brochure will be given. Patients in the laughter therapy and pursed lip breathing exercise intervention groups will be asked to perform these practices three days a week (Monday, Wednesday, Friday) for 8 weeks. At the beginning of the study, at the 4th, 8th, and 12th weeks, the Dyspnea 12-TR Scale, the COPD Evaluation Test, and the Care Dependency Scale will be administered to both the intervention and control group patients. In the application of the scales and the analysis of the data, the groups will be blinded, and the scale application will be made by an independent interviewer. After the analysis of the data in terms of normal distribution was done with the Kolmogorow Smirnov test, in the comparison of the data of the patients in the intervention and control groups; One Way Analysis of Variance or Kruskal-Wallis Analysis of Variance will be applied. Analysis of Variance in Repeated Measurements or Freidman's test will be used to calculate the change in groups over time. The statistical significance limit will be accepted as p<0.05.

DETAILED DESCRIPTION:
This research is a single-blind, randomized controlled experimental study in order to determine the effect of pursed lip breathing exercise and laughter therapy on dyspnea severity, health status and care dependence in individuals with COPD.

Research hypotheses H0-1: Pursed lip breathing exercise has no effect on the severity of dyspnea in individuals with COPD.

H0-2: Laughter therapy has no effect on the severity of dyspnea in individuals with COPD.

H0-3: Pursed lip breathing exercise has no effect on health status in individuals with COPD.

H0-4: Laughter therapy has no effect on health status in individuals with COPD. H0-5: Pursed lip breathing exercise has no effect on care dependence in individuals with COPD.

H0-6: Laughter therapy has no effect on care dependence in individuals with COPD.

Population: COPD patients receiving service in Ankara City Hospital Chest Diseases polyclinics and clinics constitute the population of the research.

Sample: Since there is no study in the literature examining the effects of pursed lip breathing exercise and laughter therapy in COPD patients, El-saidy et al. (2019) based on the study data, a sample calculation was made; Dyspnea 12 Scale scores before and after pursed lip breathing exercise (31.05± 9.2 and 22.31 ± 7.76, respectively) were found to be statistically significant (p < 0.001) (66). The effect size was calculated as 1.026 using the Priori method and the G Power program, and a total of 63 patients, at least 21 for each group, should be included in the study with a confidence interval of 95% and a power of 90%.

Research Group The patients in the institution where the study was conducted were evaluated for eligibility for the study. Voluntary consent is obtained by giving information about the research. In the study, stratified randomization method is used to ensure homogeneity between groups. Using the randomization program (https://www.randomizer.org); Stratified according to COPD Assessment Test (CAT) score (10≤ CAT≤ 25 and 25≤ CAT≤ 40) and smoking status (smoker and non-smoker); Patient lists were created as pursed lip breathing exercise intervention group, laughter therapy intervention group and control group

Research Group The patients in the institution where the study was conducted were evaluated for eligibility for the study. Voluntary consent is obtained by giving information about the research. In the study, stratified randomization method is used to ensure homogeneity between groups. Using the randomization program (https://www.randomizer.org); Stratified according to COPD Assessment Test (CAT) score (10≤ CAT≤ 25 and 25≤ CAT≤ 40) and smoking status (smoker and non-smoker); Patient lists were created as pursed lip breathing exercise intervention group, laughter therapy intervention group and control group.

The evaluation of the eligibility of the patients in the institution where the research was carried out, in line with the criteria of inclusion and exclusion from the research, is made by the thesis student. After the patient was informed about the study and their voluntary consent was obtained, the "Patient Information Form" was filled by the thesis student and according to the patient lists obtained through the https://www.randomizer.org program and stratified randomization, the patients were pursed lip breathing exercise intervention group, laughter therapy intervention group. and assigned to control groups.

Intervention Groups

Intervention Group (A):

During the first interview, the training and demonstration of pursed lip breathing exercise is performed by the thesis student in a single session, lasting approximately 40 minutes. The effects of pursed lip breathing exercise on health and its application steps are explained to the patient, and purse lip breathing exercise is performed together with the patient. In addition, the training is reinforced by giving a pursed lip breathing exercise brochure to the patient and sending a pursed lip breathing exercise application video prepared by the thesis student via whatsapp. Patients who do not have Whatsapp application are sent a video to one of their family members. After this information session, the pursed lip breathing exercise taught from the patients; They are asked to do it in their own homes, 3 days a week on Monday, Wednesday and Friday, for about 30 minutes each session, for a total of eight weeks. In order to support patients' compliance with the research; During the application process, on Mondays, Wednesdays and Fridays, the patient was contacted by the thesis student at a predetermined time, and the situation of performing pursed lip breathing exercise was questioned and recorded in the control chart . In addition, one day a week (on a day determined by the patient, Monday, Wednesday or Friday), the thesis student makes a video call to the patient on WhatsApp, and the practice of pursed lip breathing exercise is performed during the video call. After the end of the eighth week, the patients are asked to take a break from the pursed lip breathing exercise for 4 weeks (weeks 9-12), and no application is made during this period.

Intervention Group (B) During the first interview, laughter therapy training and demonstration is carried out by the thesis student in a single session, lasting approximately 50 minutes. The effects of laughter therapy on health and its application steps are explained to the patient, and the laughter therapy practice is carried out together with the patient. In addition, the training is reinforced by giving a laughter therapy training brochure to the patient and sending the laughter therapy application video prepared by the thesis student via whatsapp. Patients who do not have Whatsapp application are sent a video to one of their family members. After this information session, the laughter therapy taught from the patients; They are asked to do this in their own homes, 3 days a week on Monday, Wednesday and Friday, 30 minutes each session, for a total of eight weeks. In order to support patients' compliance with the research; During the application process, on Mondays, Wednesdays and Fridays, the patient is contacted by the thesis student at a predetermined time, and their status of doing laughter therapy is questioned and recorded in the laughter therapy application control chart. In addition, once a week (on a day determined by the patient, Monday, Wednesday or Friday), the thesis student makes a video call to the patient on WhatsApp, and laughter therapy is practiced during the video call. After the end of the eighth week, the patients are asked to take a break from the laughter therapy for 4 weeks (weeks 9-12), and no application is made during this period.

Control Group(C) Attention-match training is given to the patients in the control group. During the first interview, attention matching training is carried out by the thesis student for one time, about "Lung structure and functioning", lasting approximately 20 minutes. In addition, a brochure about lung structure and functioning is given to patients. The patients in the control group are not subjected to any other interventions throughout the study.

Data Collection The evaluation of the eligibility of the patients in the institution where the research was carried out, in line with the criteria of inclusion and exclusion from the research, is made by the thesis student. After the patient was informed about the study and their voluntary consent was obtained, the "Patient Information Form" was filled by the thesis student and according to the patient lists obtained through the https://www.randomizer.org program and stratified randomization, the patients were pursed lip breathing exercise intervention group, laughter therapy intervention group. and assigned to control groups. The scales used in the research are filled by an independent interviewer. In order to provide blinding during the data collection phase of the study, the information about which groups the patients belong to is hidden from the interviewer. In addition, patients are told not to share the information of which group they belong to during the data collection process.

Dyspnea-12 Scale, COPD Assessment Test and Care Dependence Scale 1.,2. all patients in the intervention and control groups; On the first interview day, they are told to take a break from the 4th, 8th and pursed lip breathing exercise and laughter therapy programs for 4 weeks, and they are applied again in the 12th week. The scales are filled by an independent interviewer by telephone after the completion of pursed lip breathing exercise and laughter therapy on Friday of the 4th, 8th and 12th weeks. The interviewer was given a training that included the structure, application and purpose of the scale by the thesis student.

ELIGIBILITY:
Inclusion Criteria:

* Those aged 40 and over,
* He was diagnosed with COPD as a result of medical history, physical examination and pulmonary function tests, and his CAT score is 10 and above according to the COPD Unified Assessment* of the GOLD guide; In Group B and D (1),
* There is no diagnosis of a disease that may affect the cognitive state,
* Not having a diagnosis of a physical or mental illness that will prevent communication, and able to use a telephone.
* Individuals who agree to participate in the research are included in the study

Non-Inclusion Criteria:

Those who have difficulty in verbal communication (intubation, tracheostomy, delirium, etc.)

* With a CAT score of less than 10 and in Groups A and C according to the COPD Combined Assessment* of the GOLD guide,
* Having a disorder that disrupts the cognitive process such as schizophrenia or dementia
* Alcohol, substance addiction,
* Laughter therapy was not deemed appropriate due to the diagnosis of abdominal surgery, uncontrolled hypertension, glaucoma, abdominal hernia, epilepsy in the last three months,
* Using complementary and integrative treatments such as acupuncture, meditation, yoga, massage, relaxation exercises,
* Patients who do not agree to participate in the study are excluded from the study.

Exclusion criteria

* Not complying with pursed lip breathing exercise and laughter therapy and program,
* Developing a disease that may affect the health status or a condition requiring hospitalization (COPD exacerbation, etc.) during the 12-week period during which the research will take place,
* Changes in bronchodilator and oxygen therapy regimens,
* A situation that is not suitable for laughter therapy due to the diagnosis of surgery in the abdominal region, uncontrollable hypertension, glaucoma, abdominal hernia, epilepsy,
* Patients who want to withdraw from the study are excluded from the study.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2022-08-15 (Actual); Primary Completion 2024-08-15 (Actual); Study Completion 2024-10-15 (Actual)

PRIMARY OUTCOMES:
Dyspnea in the COPD | 12 week
  Dyspnea-12 Scale, all patients in the intervention and control groups; On the first interview day, they are told to take a break from the 4th, 8th and pursed lip breathing exercise and laughter therapy programs for 4 weeks, and they are applied again in the 12th week.
  Dyspnea -12 scale, Yorke et al (2010) to measure the severity of dyspnea and to evaluate it with emotional and physical dimensions. The first 7 items measure whether the inhaled air fills all the lungs, the difficulty in breathing and the physical limitations of dyspnea in which the required effort is questioned. The other 5 items of the scale question emotional states such as stress, irritability and depression that may arise from shortness of breath. The severity of dyspnea is directly proportional to the scores obtained from the scale, and as the scores increase, the severity of dyspnea increases

SECONDARY OUTCOMES:
Health Status in The COPD | 12 week
  COPD assessment test, all patients in the intervention and control groups; On the first interview day, they are told to take a break from the 4th, 8th and pursed lip breathing exercise and laughter therapy programs for 4 weeks, and they are applied again in the 12th week.
  COPD assessment test, Jones et al. (2009) to measure health status in COPD and to evaluate the disease effect and severity. The eight-question test provides information on the grading of the disease, the scoring of symptoms, and the impact on the patient's quality of life. It covers problems such as shortness of breath, cough, and sputum production, as well as symptoms such as fatigue and sleep problems. Perfect health status: 0 points (minimum score), worst health status: 40 points (maximum score).

OTHER OUTCOMES:
Care Dependence in The COPD | 12 week
  COPD assessment test, all patients in the intervention and control groups; On the first interview day, they are told to take a break from the 4th, 8th and pursed lip breathing exercise and laughter therapy programs for 4 weeks, and they are applied again in the 12th week.
  Care Dependence Scale (CDS) Dijkstra et al. (1999) to evaluate the individual's dependence on care and to deal with addiction with its physical and psychological dimensions .The scale includes nutrition, continence, body posture, mobility, sleep, dressing, body temperature, body cleanliness, avoiding danger, verbal communication, communicating with others, worshiping, obeying rules, daily activities, recreational activities, memory and learning ability. A high scale score indicates that the patient is independent in meeting his/her care needs, while a low scale score indicates that the patient is dependent on others to meet their care needs.

CONTACTS AND LOCATIONS:
Overall Officials: Goncagul ALDAN, Principal Investigator — yüksek İhtisas University
Locations (1):
- Bilkent City Hospital, Ankara, Çamlıca Mahallesi, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data supporting the findings of this randomized controlled trial will be shared with researchers who provide a methodologically sound proposal. Data will be available upon reasonable request to the corresponding author, in accordance with ethical approval and data protection regulations.
Supporting Information: Analytic Code
Time Frame: The data will be available beginning 3 months after publication and will remain available for 2 years following publication.
Access Criteria: Access to de-identified individual participant data will be limited to researchers with an approved research proposal. Data access will be granted on a case-by-case basis and in accordance with ethical and institutional regulations.